CLINICAL TRIAL: NCT06080815
Title: Impact of Mandibular 4-Implant Overdenture Base Construction Techniques on Assessment of Occlusion With Digital Occlusion Analysis System (Within Patient Study)
Brief Title: Impact of Mandibular Overdenture Base Construction Techniques on Assessment of Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 05201021
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: According to the construction technique for the maxillary complete denture and mandibular overdentures, the patients will be classified randomly and equally into two groups.
  Group I: patients receive maxillary complete denture opposed to four implant-assisted mandibular overdenture constructed with conventional method.
  Group II: patients receive maxillary complete denture opposed to four implant-assisted mandibular overdenture constructed with CAD/CAM milling.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: patients receive maxillary complete denture opposed to conventional mandibular overdenture (Active Comparator)
  Interventions: Device: CAD/CAM Complete denture
- Group II: patients receive maxillary complete denture opposed CAD/CAM overdenture (Active Comparator)
  Interventions: Device: CAD/CAM Complete denture

INTERVENTIONS:
Device: CAD/CAM Complete denture — four implant-supported CAD/CAM complete overdenture

SUMMARY:
This within patient study will be conducted to compare between two different construction techniques (CAD-CAM Milled and Conventional techniques) of 4-implant-assisted complete mandibular overdenture bases regarding the digital occlusion force balance analysis using the OccluSense

ELIGIBILITY:
Inclusion Criteria:

* 1. Free from any systemic diseases that contraindicate dental implantation. 2. Angel's class I maxillo- mandibular relation. 3. Available inter-arch space and sufficient restorative space. 4. Nonsmokers, non-alcoholics. 5. Complaints from their conventional denture

Exclusion Criteria:

* diabetic and heavy smoker patients

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
digital occlusal analysis | 6 months
  occlusion was analyzed by occlusense device

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelghany AA, Fouad MM, Emera RMK, Askar O, Yaseen AAM. Impact of mandibular 4-implant overdenture base construction techniques on assessment of occlusion with digital occlusion analysis system (clinical crossover study). BMC Oral Health. 2025 May 30;25(1):853. doi: 10.1186/s12903-025-06228-3. PMID 40448094